CLINICAL TRIAL: NCT04073420
Title: Medtronic Cardiac Surgery Post Market Clinical Follow-up Registry
Brief Title: Medtronic Cardiac Surgery PMCF Registry
Status: Recruiting | Type: Observational
Sponsor: Medtronic Cardiac Surgery (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT18061SUR003
Record Dates: First submitted 2019-08-19; First posted 2019-08-29 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Valve Disease, Heart
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Surgical Valve Replacement and/or Repair Patients
  Interventions: Device: Surgical Heart Valve Repair Products; Device: Surgical Heart Valve Replacement Products

INTERVENTIONS:
Device: Surgical Heart Valve Repair Products — Surgical heart valve repair products.
Device: Surgical Heart Valve Replacement Products — Surgical heart valve replacement products.

SUMMARY:
This registry is being conducted to support ongoing post-market surveillance activities.

ELIGIBILITY:
Inclusion Criteria:

1. Patient or legally authorized representative provides written authorization and/or consent per institution and geographical requirements
2. Patient has or is intended to receive or be treated with an eligible product
3. Patient is within enrollment window of treatment/therapy received at the time of their initial Registry enrollment, or meets criteria for retrospective enrollment

Exclusion Criteria:

1. Patient who is, or is expected to be, inaccessible for follow-up
2. Patient prohibited from participation by local law
3. Patient is currently enrolled in or plans to enroll in any concurrent investigational drug and/or device study that may confound results

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects requiring heart valve therapy replacement and/or repair.
Sampling Method: Non-Probability Sample
Enrollment: 2700 (Estimated)
Dates: Start 2019-12-02 (Actual); Primary Completion 2039-12-31 (Estimated); Study Completion 2039-12-31 (Estimated)

PRIMARY OUTCOMES:
Identify unique failure modes | 10 years
Identify trends in adverse device effects | 10 years

CONTACTS AND LOCATIONS:
Locations (26):
- United States (11):
  - WellStar Kennestone Hospital, Marietta, Georgia
  - University of Michigan, Ann Arbor, Michigan
  - Mount Sinai Medical Center, New York, New York
  - Saint Francis Hospital, Roslyn, New York
  - Saint Josephs Hospital Health Center, Syracuse, New York
  - Duke University Medical Center, Durham, North Carolina
  - University Hospitals Cleveland, Cleveland, Ohio
  - University of Pittsburgh Medical Center UPMC Presbyterian, Pittsburgh, Pennsylvania
  - Baylor St. Luke's Medical Center, Houston, Texas
  - The Heart Hospital Plano, Plano, Texas
  - Inova, Falls Church, Virginia
- Allgemeines Krankenhaus - Universitätskliniken Wien, Vienna, Austria
- UZ Leuven, Leuven, Belgium
- Hôpital Haut-Lévêque - CHU de Bordeaux, Pessac, France
- Germany (6):
  - Schüchtermann-Klinik, Bad Rothenfelde
  - Herzzentrum Dresden GmbH Universitätsklinik, Dresden
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Albertinen-Herz- und Gefäßzentrum, Hamburg
  - Herzzentrum Leipzig, Leipzig
  - Deutsches Herzzentrum München Klinik an der TU München, München
- Onassis Cardiac Surgery Center, Athens, Greece
- Italy (2):
  - Ospedale Pasquinucci Massa, Massa
  - IRCCS Policlinico, San Donato
- Leids Universitair Medisch Centrum, Leiden, Netherlands
- Hospital Regional Universitario Carlos Haya Málaga - Hospital General, Málaga, Spain
- Inselspital - Universitätsspital Bern, Bern, Switzerland